CLINICAL TRIAL: NCT00762151
Title: Clinical Research Study to Investigate the Anti-Plaque Effect of a Prototype Toothpaste Containing an Anacor Material Via the MGMPI Method
Brief Title: A Study to Investigate the Anti-Plaque Effect of AN0128 Toothpaste
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AN0128 Periodontal Plaque
Record Dates: First submitted 2008-09-24; First posted 2008-09-30 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Dental Plaque
Keywords: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Negative Control (Placebo Comparator): Regular Toothpaste
  Interventions: Other: Negative Control (Regular Toothpaste)
- Positive Control (Active Comparator): Standard anti-plaque and anti-bacterial toothpaste.
  Interventions: Other: Positive Control (anti-plaque/anti-bacterial toothpaste)
- Prototype (Active Comparator): AN0128 Toothpaste
  Interventions: Drug: Prototype (AN0128 Toothpaste)

INTERVENTIONS:
Other: Negative Control (Regular Toothpaste) — Regular Toothpaste
  Arms: Negative Control
Other: Positive Control (anti-plaque/anti-bacterial toothpaste) — Standard anti-plaque and anti-bacterial toothpaste
  Arms: Positive Control
Drug: Prototype (AN0128 Toothpaste) — AN0128 Toothpaste
  Arms: Prototype

SUMMARY:
The objective of this study was to evaluate the anti-plaque efficacy of the Anacor prototype dentrifice as compared to commercial control products following a single use of the dentrifice.

DETAILED DESCRIPTION:
The widespread successful use of triclosan as an anti-inflammatory and anti-bacterial agent is well documented. The standard dentrifice has demonstrated a robust anti-plaque and anti-inflammatory effect providing multiple benefits. There is a clear value to identify additional agents with the same dual action with a comparable or an enhanced level of efficacy. This study examined the anti-plaque efficacy following a single use of the prototype dentifrice.

ELIGIBILITY:
Inclusion Criteria:

* Must be between ages 18 to 65 years inclusive
* Have a minimum of 16 natural uncrowned teeth (excluding 3rd molars) present
* Must give written informed consent
* Be in good general health
* Must discontinue oral hygiene for 24-hours after initial appointment
* No known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study

Exclusion Criteria:

* Medical condition which requires pre-medication prior to dental visits/procedures
* Advanced periodontal disease
* 5 or more decayed, untreated dental sites
* Diseases of the soft or hard oral tissues
* Orthodontic appliances
* Abnormal salivary function
* Use of drugs that can affect salivary flow
* Use of antibiotics one (1) month prior to or during this study
* Use of any over the counter medications other than analgesics (i.e. aspirin, ibuprofen, acetaminophen, naproxen), unless approved by the study medical staff
* Pregnant or breastfeeding
* Participation in another clinical study in the month preceding this study
* Allergic to common dentifrice ingredients
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)
* History of allergic reaction to any anti-inflammatory agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Reduction in the gingival margin plaque index in a 24-hour post-treatment (no brushing) | Baseline (time zero), 24 hour time point

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Concordia Research Laboratories, Cedar Knolls, New Jersey, United States